CLINICAL TRIAL: NCT05703165
Title: Horse-assisted Intervention and Heart Rate Variability in Participants Under Stressful Conditions
Brief Title: Horse-assisted Intervention, Heart Rate Variability & Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Baranyi, Assoc.Prof. Dr., Medical University of Graz
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 34-521
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Psychological Stress
Keywords: psychological stress; animal-assisted intervention
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- subjects with stress burden and animal-assisted intervention (Experimental): The 20-minute horse-assisted intervention takes place in compliance with basic safety precautions (safety bar between horse and participant) and after safety instruction in handling the therapy horse. The horse can be touched or stroked more or less intensively, depending on the needs and current state of mind of the study participant.
  Interventions: Behavioral: animal-assisted intervention
- subjects with stress burden and without animal-assisted intervention (Active Comparator): Study participants only observe the natural environment.
  Interventions: Behavioral: watching the countryside
- subjects without stress burden and with animal-assisted intervention (Active Comparator): The 20-minute horse-assisted intervention takes place in compliance with basic safety precautions (safety bar between horse and participant) and after safety instruction in handling the therapy horse. The horse can be touched or stroked more or less intensively, depending on the needs and current state of mind of the study participant.
  Interventions: Behavioral: animal-assisted intervention

INTERVENTIONS:
Behavioral: animal-assisted intervention — horse-assisted intervention
  Arms: subjects with stress burden and animal-assisted intervention; subjects without stress burden and with animal-assisted intervention
Behavioral: watching the countryside — just watching the countryside
  Arms: subjects with stress burden and without animal-assisted intervention

SUMMARY:
In this study, the effects of an animal-assisted intervention on people with increased stress levels are investigated. The data collected will be compared with those of participants with high stress levels but without animal-assisted intervention (participants only observe nature) and with a control group consisting of people without stress exposure.

The study will be performed in the following setting: Questionnaire examination on chronic stress, questionnaire on current well-being and heart rate variability (HRV) measurement before the horse-assisted intervention, one HRV measurement and one questionnaire examination (POMS) on current well-being after the horse-assisted intervention, one questionnaire (POMS) on current well-being 5 days after the horse-assisted intervention.

DETAILED DESCRIPTION:
The early recognition of chronic stressors, which are often neglected by those affected until physical symptoms appear, is of essential importance. In addition to psychopharmacological therapy modalities, complementary methods such as animal-assisted intervention should also be considered in order to expand the therapeutic spectrum and thus prevent stress-associated consequential harms as early as possible.

Stress has gained importance in recent years not only in the medical context, but also due to its economic relevance. Chronic stress in particular leads to numerous medically relevant secondary diseases and to increased sick leaves and even permanent incapacity to work. One possible intervention to reduce stress could be animal-assisted intervention.

Primary hypothesis: The use of animal-assisted intervention in people diagnosed with chronic stressful situations will lead to measurable increases in heart rate variability.

Secondary hypothesis: The use of animal-assisted intervention in people diagnosed with chronic stressful situations leads to improved well-being (target parameter: POMS questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Male, female and diverse
* Age between 18-75 years

Exclusion criteria:

* Animal hair allergies (especially horse hair allergies, fear of horses)
* Acute severe psychiatric conditions (e.g. psychosis)
* Persons, unable to give signed informed consent,
* All persons, who have not signed the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability | Time point 1: Baseline heart rate variability before the animal assisted intervention, Time point 2: heart rate variability immediately after the animal-assisted intervention
  Change in heart rate variability immediately after animal-assisted intervention when compared with baseline heart rate variability before the animal assisted intervention.

SECONDARY OUTCOMES:
Change in state of mood states (Profile of Mood States Questionnaire) | Time point 1: Baseline state of mood states before the animal assisted intervention, Time point 2: state of mood states immediately after the animal-assisted intervention
  Change in state of mood states immediately after animal-assisted intervention when compared with baseline state of mood states before the animal assisted intervention (Profile of Mood States Questionnaire: minimum value= -24, maximum value = 177, lower scores indicative of people with more stable mood profiles).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baranyi, Principal Investigator — Medical University of Graz, Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No